CLINICAL TRIAL: NCT05709730
Title: Follow-up of Cell Changes in the Cervix
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Joakim Dillner, Professor, Karolinska University Hospital
Other Study IDs: AGC
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Cancer of Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women aged 26-80 with atypical glandular cell (AGC) cytology result: Women in the capital region of Sweden with AGC, a concomitant human papillomavirus (HPV) analysis, and a histopathology.
  Interventions: Diagnostic Test: HPV genotyping

INTERVENTIONS:
Diagnostic Test: HPV genotyping — HPV genotyping of samples classified that were positive for "other HPV"

SUMMARY:
The purpose of the study is to follow up on cell changes detected in the cervical cancer screening program, to investigate whether they are handled with adequate quality.

DETAILED DESCRIPTION:
The aim of the study is to clarify whether follow-up of cell changes is carried out with sufficiently good quality. It is nationally recommended to perform an HPV test on mild cell changes and only refer to clinical follow-up if you are HPV positive. Descriptive statistics on HPV-testing and follow-up of quality are not available today. If HPV testing has not already been performed, archived samples with glandular cell changes will be HPV-analyzed in Cobas 4800 HPV-polymerase chain reaction (PCR), which shows data on the presence of HPV and Luminex-PCR, which shows which HPV types the samples have. Women with low-grade squamous cell changes (ASCUS and CIN1) with simultaneous HPV analysis will be followed up with data from the Swedish National Cervical Screening Registry (NKCx) from the last ten years. A register linkage with data from NKCx and the National Cancer Registry at the National Board of Health and Welfare will be carried out to determine which women have developed gynecological cancer, cervical cancer and/or pre-cancer (cancer in situ). A follow-up review of reported original cytological (cell samples) and histological (tissue samples) diagnoses will be performed by cytodiagnostics and cytopathologists, to verify the correct diagnosis.

Statistics on collection of non-organized cell samples after a partial negative sample where follow-up is not recommended are produced in aggregated form in the form of an extract from NKCx

ELIGIBILITY:
Inclusion Criteria:

* women with an AGC diagnosis between February 17, 2014 and December 31, 2018
* 23-80 years old
* resident of the Stockholm-Gotland region of Sweden

Exclusion Criteria:

-

Ages: 23 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women aged 23 years and older, residing in the Stockholm-Gotland region of Sweden who had an AGC diagnosis in a cervical cytology sample between February 17th, 2014, and December 31st, 2018. For eligibility, an HPV test result and a subsequent histopathological diagnosis is also required. HPV testing performed 40 days before or after the index sampling date is considered to indicate the HPV status of the index AGC.
Sampling Method: Probability Sample
Enrollment: 885 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
cervical intraepithelial neoplasia 3 (CIN3+) | 2014-2018
  Risk for developing CIN3+ or worse depending on HPV type

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Dillner, MD PhD, Principal Investigator — Joakim Dillner. Professor
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data available through the Swedish National Cervical Screening Registry and on request from the PI.
Time Frame: 2016-2023
Access Criteria: Ethical permission

REFERENCES:
- [Background] Norman I, Yilmaz E, Hjerpe A, Hortlund M, Elfstrom KM, Dillner J. Atypical glandular cells and development of cervical cancer: Population-based cohort study. Int J Cancer. 2022 Dec 1;151(11):2012-2019. doi: 10.1002/ijc.34242. Epub 2022 Aug 27. PMID 36029205